CLINICAL TRIAL: NCT01384136
Title: The Telomere System in Cord Blood and in the Placenta in High Risk Pregnancies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Tal Biron-Shental, Meir Medical Center, Kfar Saba, Israel
Other Study IDs: 036-2011 MMC
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Telomere Length; Mechanisms of Telomter Homeostasis; High Risk Pregnancies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High risk pregnancy
- |Control - Normal low risk pregnancies

SUMMARY:
The telomere system stabilizes the chromosomes. Telomeres are shortened during senescence, in cases of genetic instability and secondary to stress.

The investigators aim is to study the telomere system in cord blood and in the placenta immediately after the delivery in pregnancies defined as high risk pregnancies following sterss events such as placental insufficiency, preeclampsia, diabetes.

The investigators intend to compare the telomere system in maternal blood to cord blood and to placental biopsies and to study the influence of different stressogenes on this system.

ELIGIBILITY:
Inclusion Criteria:

* Third trimester post delivery
* Intrauterine growth restriction
* Preeclampsia
* Diabetes
* Control - low risk normal pregnancies

Exclusion Criteria:

* Patients who do not want to participate
* Known HIV or Hepatitis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: High risk pregnancies, third trimester, after the delivery/
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel